**Title:** Adapting Diet and Action for Everyone (ADAPT+) Study Protocol and Statistical Analysis Plan.

# NCT04800432

**Last updated:** 11/19/2021

Study Title: ADAPT+: Optimizing an Intervention to Promote Healthy Behaviors in Rural, Latino Youth with Obesity and their Parents, using Mindfulness Strategies.

Proposal # #Pro00039979

PI: Marilyn Stern, Ph.D.

Dept. of Child and Family Studies

Guidelines for studies meeting the criteria for expedited or full Board review:

#### A. Overview:

1. Rationale for the study, area of current scientific concern and why the research is needed;

Rates of obesity among Latino youth is increasing exponentially.<sup>1-4</sup> It is estimated that unless this trend is reversed, 90% of US-born children of Mexican immigrants will be of overweight or obese status by 2030,<sup>5</sup> particularly those living in rural communities.<sup>6-10</sup> With a rise in obesity, Latino youth are at increased risk for metabolic syndrome, type 2 diabetes, cardiovascular disease and cancer.<sup>11-14</sup> Lifestyle interventions have predominantly depended on education and cognitive-behavioral strategies to improve diet and physical activity (PA), with parent- focused interventions showing the most consistent success for youth.<sup>15,16</sup> Still, these studies often produce only modest and short-term results.<sup>17</sup> The link between parent stress and offspring obesity has been shown,<sup>18</sup> yet the role of parent stress on obesity has not been well addressed in interventions for reducing obesity in Latino youth. Evidence implicates stress in disordered eating and obesity<sup>21,22</sup> and parent stress relates to risk factors for childhood obesity.<sup>18</sup> Mindfulness-based programs are successfully delivered to low-income, minority, public school students;<sup>23</sup> however, few studies target Latino families.

2. Living in a rural community compounds the health care disparity of Latino youth and obesity.

Most Latinos in Florida (outside of Miami) live in rural areas and work as migrant farmworkers. <sup>10,32</sup> Latino youth living in rural areas are 25% more likely to have overweight/obesity than Latinos in urban areas. <sup>7,10</sup> Compared with Latinos living in urban areas, Latinos in rural areas typically consume more meals with friends and relatives outside the home, making food choices more difficult. Lack of access to affordable, healthy foods; few community resources; acculturation-related dietary changes (e.g., eating more processed and fast foods<sup>31</sup>) and poverty are key contributing factors to obesity. <sup>7-9</sup> Children in households living below the poverty line have 243% higher odds of developing childhood obesity than children living above the poverty threshold. <sup>10,32,33</sup> Latino rural communities have been largely ignored despite the rising economic, social, and personal burden of obesity, including medical care costs. <sup>34,35</sup>

3. Link between Latino parent stress and offspring obesity.

A growing body of evidence implicates stress in obesity, <sup>21,22</sup> especially related to food choices and preferences. <sup>36</sup> An American Psychological Association survey reported 39% of adults overeat or increase intake of calorie-dense foods in response to stress. <sup>21</sup> Moreover, inability to maintain improvements in healthy lifestyle behaviors is linked with psychological distress in individuals with obesity. <sup>37</sup> In youth, chronic stress has been linked with larger waist circumference and BMI. <sup>38</sup> Latino families are especially subject to specific and burdensome stressors (e.g. economic hardship and fear of family member deportation) that may predispose them to behaviors that increase obesity. The large scale "SOL" investigation of Latino youth and their caregivers (n=473; children aged 8–16 years) found the incidence of youth obesity

increased substantially with the number of caregiver stressors. <sup>18</sup> Long work hours, common among migrant worker families, can reduce parent involvement, including uninvolved feeding style, which can increase risk of obesity in youths. <sup>39,40</sup> Specifically, parent stress is associated with decreased physical activity (PA), overeating <sup>41</sup> and higher body weight in both children and parents. <sup>42</sup> Given the literature that highlights the importance of focusing on parents in changing eating, PA and other health behaviors in youth, targeting parent stress to impact these behaviors may be key. <sup>15,16</sup> However, there is a lack of culturally competent, evidence-based, interventions to address stress and its concomitant relation with the urgent public health issue of overweight/obesity among rural Latino youth. <sup>35</sup>

# 4. Critical barriers to progress in the field:

Most obesity interventions for Latino youth report mixed findings, are small in scope and exploratory <sup>28,43,44</sup> and fail to incorporate key factors important for Latinos living in rural communities. 17,31,44,45 For example, community-based interventions promote better 'buy-in' from Latino families, <sup>17,28,44</sup> particularly utilization of promotoras (community health workers), <sup>29</sup> yet most available studies have not delivered interventions in a community setting. 46 Moreover, the "state of the obesity intervention field" suggests that interventions that are parent-focused, but also involve the entire family, show the most promise. 16 This is particularly the case in Latino families because of the strong commitment to the family system ("familismo"), yet most extant studies involving Latinos do not include children. The majority of studies also have lacked: rigorous experimental methodology, manualized treatment programs that measure both physical activity (PA) and eating behaviors, culturally appropriate strategies, <sup>31,44,45</sup> and longitudinal follow-up assessments. <sup>17</sup> To date, obesity interventions with Latinos have also lacked sufficient attention to barriers to success, including acculturation considerations which include, dietary changes such as, using larger quantities of sodium, oils, and sugars; consuming an excess of sugar-sweetened beverages and fast food; and having a suboptimal consumption of fruits and vegetables. 17,48-56 We argue here that mixed results of interventions may also be due to their failure to successfully address multi-faceted psychosocial risk factors, such as parent stress.<sup>57</sup> Multifaceted approaches must be taken into consideration in designing intervention strategies to increase the effectiveness and sustainability of health behavior changes for migrant Latino families. In response to these barriers to success, our refined intervention will focus not only on acculturation considerations of dietary changes, PA, but also parent stress within the family.

### The research questions, objectives and purpose;

The purpose of this study is to refine and optimize an obesity intervention with rural underserved Latino children and their parents that combines a standard family-based behavioral approach, the "gold standard" for pediatric obesity treatment, <sup>16,47,77,78</sup> with a mindfulness approach focusing on stress reduction (now ADAPT+).

Aim 1: Refinement of and optimization of ADAPT+ (ADAPT + mindfulness parent stress reduction combination) manual and intervention.

We assess acceptability of ADAPT and the integration of mindful parenting stress reduction (ADAPT+) to increase healthy lifestyle behaviors consistent with the needs of Latinos living in rural communities. We will conduct a series of focus groups: 1) with our community health facilitators/promotoras. Promotoras are community members who have been acculturated in the US but retain credibility with the target population.<sup>28,29</sup> 2) a series of focus groups with parents

of children (8-12 years old) with obesity to obtain feedback and to refine each of our 6 integrated sessions and evaluate optimization of ADAPT+ sessions.

Aim 2: A small, randomized feasibility and acceptability study (ADAPT+ vs. Enhanced Usual Care comparison/EUC).

Aim 2 will be conducted in two rural communities. This aim evaluates: study sample selection and recruitment, willingness to be randomized and retention; fidelity of intervention administration, intervention adherence, and further refinement of manuals, feasibility of data collection procedures, including collecting a battery of measures from parents and children,\* data quality and sensitivity of our measures to our intervention effects over time – from baseline, post-intervention (after 6 sessions), and then 3-months post-intervention. We anticipate that compared to EUC, parent-child dyads in ADAPT+ will have a lower attrition rate and will report greater program satisfaction, and our eating, PA and stress-related measures will be sensitive to the intervention.

The foundation/basis of the proposed study is that parent stress reduction via mindfulness strategies will increase access to mind-body practices that may support and promote implementation of healthy behaviors in both parents and children. This project will provide crucial data to inform a larger trial application to test whether adding mindfulness techniques increases the ability of parents to assist their children in keeping healthy behaviors related to eating and physical activity. This programmatic research advances the understanding of mechanisms of behavioral interventions for improving health and well-being using mind-body practices.

#### B. \*Measures to be used:

Baseline, post-intervention and 3-months follow-up:

<u>Child BMI</u>: Height (to the nearest 1/4 inch) using a stadiometer and weight (to the nearest 1/4 pound) using a medical balance beam scale will be measured by study staff. The CDC Growth Charts will be used to obtain the continuous child BMI z score for gender and age. Our nurse scholar and RNP co-I completes all the anthropometric assessments.

<u>Child Waist-to-Hip Ratio:</u> Circumference of the hip (girth of hips above the gluteal fold) and waist (narrowest part of torso above the umbilicus and below the xiphoid process) will be measured by study staff using an anthropometric measuring tape and used to calculate continuous Waist-to-Hip Ratio. Our nurse scholar and RNP co-I completes all the anthropometric assessments.

Resting Blood pressure for children: assessed in triplicate using an automated blood pressure analyzer, with the participant in a seated position. Elevated BP is defined as either systolic or diastolic BP >90th%ile for age, sex, and height. Our nurse scholar and RNP co-I completes all the anthropometric assessments.

<u>Child Food and Physical Activity Questionnaire</u>: The questionnaire consists of 11 questions on food and physical activity behaviors for youth participants in the study. This was adapted from the USDA Youth Expanded Food and Nutrition Education Program (EFNEP) evaluation tool, the EFNEP 3rd-5th Grade Survey, which was designed and tested by Purdue University Extension Program.

<u>Parent BMI</u>: Height (to the nearest 1/4 inch) using a stadiometer and weight (to the nearest 1/4 pound) using a medical balance beam scale will be measured by the study staff and used to calculate continuous adult BMI score. Our nurse scholar and RNP co-I completes all the anthropometric assessments.

<u>Parent Waist-to-Hip Ratio</u>: Circumference of the hip (girth of hips above the gluteal fold) and waist (narrowest part of torso above the umbilicus and below the xiphoid process) will be measured by the study staff using an anthropometric measuring tape and used to calculate continuous Waist-to-Hip Ratio. Our nurse scholar and RNP co-I completes all the anthropometric assessments.

<u>Resting Blood pressure for Parents</u>: assessed in triplicate using an automated blood pressure analyzer, with the participant in a seated position. Elevated BP is defined as either systolic or diastolic BP >90th%ile for age, sex, and height.

Our nurse scholar and RNP co-I completes all the anthropometric assessments.

<u>Dietary Habits</u>: The Latino Dietary Behaviors Questionnaire: This 13-item self-report survey of dietary habits (in Spanish) assesses 4 areas of eating behavior -- healthy dietary changes; types of drinks consumed, number of meals per day and fat consumption. The LDBQ factor structure is relatively stable over time, and correlates significantly with the 24-HR dietary recall measure and clinical variables such as BMI, and behavioral indicators of diet. It is specifically designed for low literacy populations and has been validated in large samples of ethnically diverse Spanish speaking samples.

<u>Perceived Stress Scale (PSS)</u>: Parents complete the 14 item self-report scale that asks participants about their feelings in the past month. The PSS measures psychological stress associated with sex, age, education, income, employment status, and a number of other demographics.

Mindful Eating Questionnaire (MEQ): Parents will complete the Recognize Subscale of the MEQ. The MEQ is a 28-item scale developed to measure the construct of mindful eating, a nonjudgmental awareness of the physical and emotional sensations associated with eating. The Recognize subscale has 9 items and is designed to assess an individual's ability to stop eating when full.

At <u>Baseline Only</u>: Parents will complete the <u>Stephenson Multigroup Acculturation Scale (SMAS)</u>, and a short demographic questionnaire.

Exit survey: At the end of the intervention, after 6-weeks, parents in both conditions will complete a brief exit survey to assess their overall satisfaction with the intervention and their opinion of its impact on their knowledge of childhood obesity and healthy eating, physical activity behaviors, mindfulness parent stress reduction approaches, as well as how well the content fit their needs and cultural values. For example, what they liked/disliked about the intervention, what additional information they might have wanted, the extent to which they felt they increased their understanding of healthy lifestyle behaviors and stress reduction strategies.

#### C. Study Design:

1. The study design including information that is needed to answer the research questions;

The study design proposes a refinement and optimization of the original ADAPT obesity intervention protocol to include mindfulness parent stress reduction strategies (ADAPT+),

setting the basis for an efficacy trial of ADAPT+'s efficacy for improving Latino families' eating and PA behaviors.

Targeting two health care disparities by developing a culturally relevant obesity intervention for high-risk Latino youth and their parents (ethnic minorities) living in rural communities (a geographic health disparity). We synthesize behavioral family-based obesity interventions with culture-specific components to promote adaptive health behaviors in a high-risk and underserved population.

Incorporating mindfulness parent stress reduction strategies into a behavioral healthy lifestyle program. Mindfulness-based approaches are shown to decrease stress and contribute to improved eating and PA behaviors, supporting our inclusion of a mindfulness component. This project is the first to incorporate mindfulness to potentially enhance initial and sustained weight loss among Latino youth.

Incorporating bilingual community liaisons from the same community as participants will increase potential for program dissemination, as well as participant engagement. This study will integrate bilingual promotoras from the same community as participants as intervention facilitators.

Individualizing behavior change goals is expected to increase families' commitment to and engagement in working toward their weight-related health goals.

Using a multi-family format, which is consistent with community and collectivist Latino family values. Mutual support within and across child/parent pairs is likely to promote engagement.

Partnering with an established and respected community-based organization, the Hispanic Services Council (HSC). HSC shares a mission consistent with our aims: the reduction of health and education disparities in Latino families. This partnership is expected to increase project buyin of Latino migrant families and contribute to the dissemination of the program.

### 2. Sample size;

For Aim 1a: we will conduct a focus group with 6 promotoras (community health workers)

For Aim 1b: we will conduct two focus groups with a total of 20 (max) Latina mothers of 8- to 12-year-old children who are overweight or obese (85<sup>th</sup> BMI percentile)

For Aim 1c: we will conduct focus groups using one cohort of mothers and their children meeting eligibility to further refine the ADAPT manual. Parents and children will attend all six sessions of ADAPT+ sessions and provide feedback for manual optimization. Latina meal preparers in the family (primarily mothers) and their 8- to 12-year-old children (up to 10 children) will participate.

Summary of Participants 6 community health workers (promotoras or group facilitators); 30 Latina mothers (Aims 1a and b) 10 children (Aim 1c); <u>Total = up to 46 participants</u> (non-clinical trial portions of the project)/

Aim 2: A small pilot RCT will be conducted (clinical trial). There will be cohorts of 8-10 child/parent pairs at each site (2 sites), and 3 intervention cycles. Estimating that all cohorts are the minimum of 8 pairs, we will have a total minimum target sample size of 48 pairs, or 96 total participants (48 parents and 48 youth). If all groups are the maximum of 10 pairs, we will have a maximum total sample size of 60 pairs, or 120 total participants (60 parents and 60 youth). We

aim for a minimum of 48 pairs with a possible range of 48 to 60 pairs based on our study design. Starting in Year 2, in total we will run 3 ADAPT+ and 3 EUC cohorts.

# D. Study Population inclusion and exclusion criteria;

- C.3.2. Eligibility criteria. Promotoras trained to conduct focus groups by our study site partner, HSC, will identify families living in our target community meeting our eligibility criteria:
- 1. Latino families with a child between the ages of 8 and 12; Note: pre-adolescents are targeted as this is a developmentally critical age group in terms of developing health-behavior skills and is an age group identified as in need of further study in the Latino population. 2. Child with a BMI %ile of 85 or higher; and 3. The target parent is at least 18 years old, is the main meal preparer, speaks and reads Spanish at a minimum of a 4th grade reading level (able to follow basic instructions in Spanish), and able to perform simple physical exercises. Although both parents and/or other caregivers can participate in the group, only data from the primary parent (main meal preparer) will be used for analyses. The parent is ineligible if he/she is non-ambulatory, is pregnant, or has a medical condition that may be negatively impacted by PA. A child who has a medical/developmental condition that precludes weight loss using conventional diet and PA methods or has been on antibiotics or steroids in the previous three months is also ineligible.

### E. The expected results of the research, such as reports, papers, and contributions to theory;

We posit that mindfulness can improve intervention engagement (increasing receptiveness), which are demonstrated critical barriers to Latino families participating in childhood obesity interventions, by simultaneously reducing stress and enhancing the learning process around eating and PA. ADAPT plus mindfulness parent stress reduction to increase healthy eating and PA lifestyle behaviors in both parents and their children.

### F. Name of the Principal Investigator and Faculty Advisor if applicable;

Dr. Marilyn Stern

### G. Any potential risks to the subjects;

This research is considered to be minimal risk. That means that the risks associated with this study are the same as what the participant would face every day. There are no known additional risks to those who take part in this study.

#### H. Any experimental procedures or interventions that will be implemented;

The study will assess acceptability of the integration of mindfulness parenting stress reduction into Adaptando Dieta y Acción Para Todos (ADAPT) to increase healthy lifestyle behaviors by: conducting a series of focus groups with our community health facilitators/ promotoras and parents of children (8-12 years old) with obesity to obtain feedback about and refine each of our 6 integrated sessions and evaluate optimization of ADAPT+ sessions.

More specifically, aim 1A) In-depth focus groups with promotoras (3 promotoras from each of our 2 target communities). These groups will be led by Stern and Redwine, and a bilingual

research assistant (RA) to elicit promotoras' impressions and obtain feedback about our proposed 6-session program, ADAPT+. Each proposed component of the program will be reviewed and feedback will be elicited from participants. Aim 1B) Two iterative one-session focus groups of parents (6-10 parents in each group) of children with obesity between the ages of 8 and 12 will be conducted. The ADAPT+ intervention manual will be examined and modified accordingly with each two-hour focus group iteration led by trained promotoras from the same community as participants, along with bilingual RAs to maintain focus group fidelity (e.g., detailed note taking). As they have done in past focus group research promotoras will be trained to elicit feedback via structured interviews and prompts on each of our eight sessions of our combined ADAPT+ intervention manual, including session goals and activities, and their relevance. We are particularly interested in the acceptability (e.g. cultural and individual) of the mindfulness parent stress reduction components, and how best to integrate them into our manualized ADAPT program. In the second group led by promotoras, parents will be asked to provide us with feedback about our refined ADAPT+ manual based on the modifications made after the first parent focus group. Our trained RAs will also use cognitive interviewing strategies to elicit specific feedback from individual parents to help with the further refinement of the ADAPT+ manual. All focus group sessions and interviews will be audiotaped for later coding.

Aim 1C is to further refine ADAPT+ by recruiting a third group of 8-10 primary meal preparers from one of our target communities meeting our eligibility criteria. Children of these parents will also participate in a parallel program at the same time, but separately. For Aim 1C, we will have two of our trained promotoras conduct the revised ADAPT+ 6 sessions intervention in Spanish to parents so that we obtain further information to optimize our ADAPT+ manual.

For Aim 2, the same procedures will be used for recruitment as for Aim 1, but groups of families, or cohorts, during each intervention cycle will be assigned to either ADAPT+ or EUC in line with the following procedures: The ordering of which community site (Plant City or Wimauma) offers ADAPT+ first will be randomly selected for cycle 1, with one community site offering ADAPT+ and the second community site offering EUC. Cycle 2 will counterbalance cycle 1, with the community site that offered EUC in cycle 1 now offering ADAPT+ in cycle 2. ADAPT+ will be randomly assigned to a community site again in cycle 3, with the second community site offering EUC (see Table 3 below). At the baseline session, our bilingual study staff member/RA will answer questions and get parental signed consents and children's verbal assents. The study staff member, along with our co-I Dr. Rodriguez (a certified RNP), will then conduct all anthropometric, stress-related and behavioral assessments.

| Table 3. Hypoth | Table 3. Hypothetical Counterbalance Design | |
|---|---|---|
| | Dover Clinic | Wimauma Clinic |
| Cycle 1 | ADAPT+ Cohort 1 | EUC Cohort 1 |
| Cycle 2 | EUC Cohort 2 | ADAPT+ Cohort 2 |
| Cycle 3 | ADAPT+ Cohort 3 | EUC Cohort 3 |

# Summary of the ADAPT+ sessions

| | le 2. Session Content of Mindfulness parent stress reduction + A | DAPT | |
|---|---|---|---|
| | te: all sessions include Home Practice suggestions | | |
| Sess | ion 1: Overview & Get Ready for Success | Session 2: Mindful Meal Prep | |
| | <ol> <li>Introductions (8 minutes)</li> <li>Health risks of obesity in Latino families</li> </ol> | <ol> <li>Homework review and raffle for goal settin<br/>(quickly review barriers) (10 minutes)</li> </ol> | ıg |
| | a. BMI charts review for parents and children (10 | 2. Mindful moment (3 minutes) | |
| | minutes) | 3. Reading labels in English (20 minutes) | |
| | b. Challenges of living in rural area and | 4. Portion Sizes | |
| | acculturation (adaptation to culture; foods, etc.) | a. Determining portion sizes (2 mi | nutes) |
| | (5 minutes) | <ul> <li>b. MyPlate. Culturally tailored stra</li> </ul> | ategies |
| | 3. Effects of Stress on health (10 minutes) | for portion control (10 minutes) | |
| | Connection between parents feeling stress and | c. Limiting portion sizes (10 minu | |
| | effects on their children (5 minutes) | d. Don't drink your calories (5 mir | nutes) |
| | 4. Practicing mindfulness (1 minute) a. Mindful stretching/moving (5 minutes) | <ol> <li>High risk eating situations (10 minutes)</li> <li>a. Mindful eating during social large</li> </ol> | *** |
| | b. Short mindful eating exercise (5 minutes) | gatherings (1 minute) | ge |
| | 5. Eating healthy | b. Hunger Scale (5 minutes) | |
| | a. Reading labels (5 minutes) | c. S.T.O.P (5-8 minutes) | |
| | b. Determining portion sizes (2 minutes) | d. Body scan (8 minutes) | |
| | 6. Creating SMART goals (8 minutes) | <ol><li>Joint Goal Setting and home practice instru</li></ol> | ctions |
| | 7. Joint Goal Setting and home practice instructions (10) | (10 minutes) | |
| | <ol> <li>Goal Setting (Mindful eating home practice)</li> </ol> | a. Goal setting (PA and healthy ea | |
| | | Goals, start small and increase of | over |
| | | time) | |
| Soco | ion 3: Parenting in the moment & Increasing Healthy | b. S.T.O.P home practice Session 4: Mindfulness and Making Healthy Behav. | ior |
| | styles | Choices + Get Moving! | 101 |
| Liic | Homework review and raffle for goal setting (5 minutes) | Homework review and raffle for goal setting | ıg (5 |
| | 2. Mindful moment (3 minutes) | minutes) | 5 (- |
| | 3. Culturally tailored ways to meal planning | <ol><li>Mindful moment (3 minutes)</li></ol> | |
| | <ol> <li>Meal Skipping and Meal Planning.</li> </ol> | <ol><li>Effects of sedentary lifestyles (10 minutes)</li></ol> | |
| | b. Eating on a budget. | a. Impact of screen time | |
| | c. Breakfast is for the Brain. | 4. Being healthy & PA (25 minutes) | <i>(</i> * |
| | d. Learn to like it. 4. Parenting and role modeling (20 minutes) | Making healthy behavior choice mindful walking, dancing, exerc | |
| | a. Parental styles | at home) | Jishig |
| | b. What is role-modeling? (10 minutes) | b. Scheduling physical activity | |
| | c. Guild, parenting, and mindfulness | c. Screen-free activities (handout) | |
| | 5. Managing stress. Reacting vs responding: | <li>d. Time management and exercise</li> | (10 |
| | <ol> <li>Parents replenish their inner resources.</li> </ol> | minutes) | |
| | b. Mindful communication. | e. Sleep hygiene | |
| | c. Non-judging. | 5. Dealing with stress using mindfulness and | PA |
| | d. Seated meditation (Awareness of breath and thoughts; 8 minutes) | (including the family in activities) a. Being present and in the momer | at. |
| | 6. Joint Goal setting and home practice instructions | b. Mindful stretching/moving (8 | π. |
| | a. Goal setting (PA and healthy eating Goals, | minues). | |
| | parents' role-modeling) | 6. Joint Goal setting and home practice instruc | ctions |
| | <ul> <li>Body scan at bedtime home practice and</li> </ul> | <ul> <li>Goal setting (PA and healthy ea</li> </ul> | ting |
| | mindful listening | Goals) | |
| | | <ul> <li>b. Mindful walking home practice</li> </ul> | |
| | ion 5: Mindful Eating + Observing vs. Judging | Session 6: Practice not Perfection + | |
| 1) 2) | Homework review and raffle for goal setting | Progress & Dealing with Setbacks | |
| 3) | Mindful moment (3 minutes) Food accessibility | Homework review and raffle for goal setting | |
| 4) | Making favorite dishes healthier (e.g., tortillas) | a) Overcoming barriers (difficulties in meal | |
| ., | a) Food label activity for usual foods. | planning) | |
| | b) Increase intake of fruits and vegetables. | 2) Mindful moment (3 minutes) | |
| 5) | Examining & changing hunger cues | Progress discussion | |
| | a) S.T.O.P (3 minutes) | 4) <u>Body scan (8 minutes)</u> | |
| | i) Revisit hunger scale if necessary | 5) Practical suggestions for continuing progress | |
| | b) Mindful eating exercise (observing/letting go of judgements; 8 minutes) | <ul> <li>a) Review the healthy recipes book (and may)</li> </ul> | be |
| 6) | Mindfulness, stress and stress reactivity | potluck). | |
| , , | a) Implementing mindfulness in daily life. Barriers and | <ul> <li>b) Coping with setbacks to healthy eating, PA</li> </ul> | . & |
| | facilitators to mindfulness | mindfulness goals in the long-term. | |
| 7) | Joint Goal setting and home practice instructions | | |
| l . | a) Goal setting (PA and healthy eating Goals/meal planning, | | |
| | increase fruit/vegetable intake in meal planning) | | |
| | b) S.T.O.P home practice during a stress-evoking situation at | | |
| | home | | |

Each session begins with a review of the previous week, monitoring of goal progress, and reviews of weekly family meals. A range of exercises and activities are included in each session. As indicated in Table, several sessions focus on diet and preparing easy, practical meals. Foods discussed include those common within this culture and healthy adaptations, as appropriate. ADAPT+ also includes an emphasis on increasing PA for the whole family. This will be

achieved via guided goal setting and self-monitoring. The mindfulness parent stress reduction approach is based on stress reduction methods by Kabat-Zinn and mindful eating and awareness of family choices. The content includes cultivating mindfulness, such as present-focused awareness, non-judgment of inner experience, nonreactivity to experience, and cultivating compassion, particularly in family lifestyle choices. Sessions include, 1) Mindfulness based stress reduction overview; 2) Mindful Meal Preparation; 3) Parenting in the moment and increasing healthy lifestyles; 4) Mindfulness and making healthy behavior choices; 5) Mindful eating; Observing vs Judging; 6) Practice not perfection.

# I. Any potential benefits to subjects;

There is no guarantee of direct benefits by taking part in this research study. This study will increase awareness of how to improve a healthy lifestyle program for Latino families in rural areas and how to work with these families to help them develop a healthy lifestyle.

### J. Compensation

For Aim 1c parents will be compensated with a \$20 gift card after the first assessment session and a fitness tracker after the last assessment session. Participating children will also receive a fitness tracker and may get some small prizes for their participation throughout the project (e.g., colorful beads).

For Aim 2 parents will be compensated with a \$10 gift card after the first session, a \$20 gift card for completing the post-intervention exit survey assessment after the 6-weeks of the program, and a \$25 gift card for completing the 3-months follow-up measures.

Human subjects considerations including description of the informed consent process; if applicable include a discussion of safeguards that are in place to protect potentially vulnerable subjects such as children, prisoners, the cognitively impaired, institutionalized or critically/terminally ill; discussion of how the privacy and confidentiality of the subjects will be maintained

Consent and assent will be obtained by a bilingual research assistant. Consent forms will be available in both English and Spanish. Parents may choose their preference. Consent forms will be written in at a fourth-grade level. Reading at this level has been made part of the inclusion criteria. Parents will also be briefed on the study before signing consent forms and are free to ask questions. Children will get all the information explained using a children friendly language and verbal assent will be requested.

Due to Covid-19 consent process for Aim 1B will be slightly different than originally planned. For this Aim, our promotoras (community health workers) will be running small focus groups in person, with appropriate precautions, social distancing, and masks, as previously approved. However, it is likely that our bilingual research assistants (RA) will only participate via videoconferencing, following USF safety standards. For this reason, informed consent from these mothers will be acquired via videoconferencing. Mothers will have written copies of the consent forms (approved in 5/23/2019) and our RA will go over the consent via videoconferencing and then have each mother sign the consent form prior to beginning the focus group with the promotoras. These consent forms will then be collected and mailed back to USF in a secure envelope to be stored in our locked file cabinet. We will provide the Hispanic Services Council director with these envelopes and gift cards for participants prior to the focus groups being

scheduled. The RA will then continue to monitor the focus groups, as originally planned, via videoconferencing.

To protect confidentiality, personal information will be restricted to the research team, government or university individuals who need to know about the study, and the USF Institutional Review Board. Any information that is published will not contain names or other identifiable information. Data will be restricted to the research team and any physical records will be locked away. Participants will not be provided any identifiable information about individuals other than themselves. Lastly, we will not receive or disclose any protected health information.

### K. Statistical Analysis Plan

Preliminary evaluation of participants' response to the interventions will be examined using quantitative data. While evaluation of outcomes is more appropriate for a fully-powered R01, we will examine variance and effect sizes of key outcomes from pre- to post-intervention, as well as post-intervention to 3-month follow-up using non-parametric tests and confidence intervals. The randomized trial is powered to detect an average estimated effect size equivalent to Cohen's d of 0.50 with the minimum sample size of 96 participants (i.e., 48 children, 48 parents). Analyses will explore potential patterns related to attrition. Every effort will be made to collect follow-up data from all participants, regardless of whether they completed the intervention.

### L. Research references:

- 1. Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. Jama. 2014;311(8):806-814.
- 2. Houston K, Waldrop JB, R M. Evidence to guide feeding practices for Latino children. J Nurse Pract. 2011;7:271-276.
- 3. Lichter DT. Immigration and the New Racial Diversity in Rural America. Rural Sociol. 2012;77(1):3-35.
- 4. Bates LM, Acevedo-Garcia D, Alegria M, Krieger N. Immigration and generational trends in body mass index and obesity in the United States: results of the National Latino and Asian American Survey, 2002-2003. Am J Public Health. 2008;98(1):70-77.
- 5. Tuñón-Pablos E, J D. Risk Factors for Overweight and Obesity among Mexican Children in New York. International Journal of Population Research. 2016.
- 6. Haldeman CJ, Giles WH, Rashidee A. Hospitalization of patients with heart failure: National Hospital Discharge Survey, 1985 to 1995. Am Heart J. 1999;137(2):352-360.
- 7. Lutfiyya MN, Lipsky MS, Wisdom-Behounek J, Inpanbutr-Martinkus M. Is rural residency a risk factor for overweight and obesity for U.S. children? Obesity (Silver Spring, Md). 2007;15(9):2348-2356.
- 8. Jilcott SB, Wade S, McGuirt JT, Wu Q, Lazorick S, Moore JB. The association between the food environment and weight status among eastern North Carolina youth. Public Health Nutr. 2011;14(9):1610-1617.
- 9. Rodriguez R, Weffer SE, Romo J, Aleman A, Ortiz RM. Reduced physical activity levels associated with obesity in rural Hispanic adolescent females. Childhood obesity (Print). 2011;7(3):194-205.
- 10. Florida Department of Health. Population by year by county. In: Florida population estimates [2008-2013], ed. Tallahassee, FL: Florida Department of Health. [Table generated by active query]. www.floridacharts.com/FLQUERY/Population/PopulationRpt.aspx; 2015.
- 11. Wang Y, Beydoun MA. The obesity epidemic in the United States--gender, age, socioeconomic, racial/ethnic, and geographic characteristics: a systematic review and meta-regression analysis. Epidemiol Rev. 2007;29:6-28.
- 12. Butte NF, Cai G, Cole SA, Comuzzie AG. Viva la Familia Study: genetic and environmental contributions to childhood obesity and its comorbidities in the Hispanic population. Am J Clin Nutr. 2006;84(3):646-654; quiz 673-644.
- 13. Stovitz SD, Schwimmer JB, Martinez H, Story MT. Pediatric obesity: the unique issues in Latino-American male youth. Am J Prev Med. 2008;34(2):153-160.
- 14. Wenten M, Gilliland FD, Baumgartner K, Samet JM. Associations of weight, weight change, and body mass with breast cancer risk in Hispanic and non-Hispanic white women. Ann Epidemiol. 2002;12(6):435-434.
- 15. Golan M, Crow S. Targeting parents exclusively in the treatment of childhood obesity: long-term results. Obes Res. 2004;12(2):357-361.

- 16. Janicke DM, Steele RG, Gayes LA, et al. Systematic review and meta-analysis of comprehensive behavioral family lifestyle interventions addressing pediatric obesity. J Pediatr Psychol. 2014;39(8):809-825.
- 17. Leung, MM, Cavalcanti, OB, El Dada, A, Brown, M, Mateo, MF, Yeh MC. Treating Obesity in Latino Children: A Systematic Review of Current Interventions. International Journal of Child Health and Nutrition. 2017;6(1):1-15.
- 18. Isasi CR, Hua S, Jung M, et al. The Association of Parental/Caregiver Chronic Stress with Youth Obesity: Findings from the Study of Latino Youth and the Hispanic Community Health Study/Study of Latinos Sociocultural Ancillary Study. Childhood obesity (Print). 2017;13(4):251-258.
- 19. Stern M, Lescano, C., Lopez Castillo, H., Lynn, C., & Bleck, J. Adaptando Dieta y Accion Para Todos (ADAPT): Targeting diet and physical activity of Latinos living in rural communities in Florida. In I. B. Thurston (chair). Culturally Responsive Assessments and Interventions to Address Pediatric Obesity: A Collaborative Symposium of the Diversity and Obesity SIGs. Society of Pediatric Psychology; 2017; Portland, OR.
- 20. Stern M, Redwine, LS, Rancourt D, Rodriguez, C, Castillo, H, Lescano, C. Developing Adaptando Dieta y Acción Para Todos (ADAPT): Improving healthy lifestyles among Latino parents and children living in a rural community. (submitted for publication). 2019.
- 21. Tsenkova V, Boylan JM, Ryff C. Stress eating and health. Findings from MIDUS, a national study of US adults. Appetite. 2013;69:151-155.
- 22. Block JP, He Y, Zaslavsky AM, Ding L, Ayanian JZ. Psychosocial stress and change in weight among US adults. Am J Epidemiol. 2009;170(2):181-192.
- 23. Daly P, Pace T, Berg J, Menon U, Szalacha LA. A mindful eating intervention: A theory-guided randomized anti-obesity feasibility study with adolescent Latino females. Complement Ther Med. 2016;28:22-28.
- 24. Black DS, Fernando R. Mindfulness Training and Classroom Behavior Among Lower-Income and Ethnic Minority Elementary School Children. Journal of child and family studies. 2014;23(7):1242-1246.
- 25. Dalen J, Brody JL, Staples JK, Sedillo D. A Conceptual Framework for the Expansion of Behavioral Interventions for Youth Obesity: A Family-Based Mindful Eating Approach. Childhood obesity (Print). 2015;11(5):577-584.
- 26. Onken LS, Carroll KM, Shoham V, Cuthbert BN, Riddle M. Reenvisioning Clinical Science: Unifying the Discipline to Improve the Public Health. Clin Psychol Sci. 2014;2(1):22-34.
- 27. Naar S, Czajkowski SM, Spring B. Innovative study designs and methods for optimizing and implementing behavioral interventions to improve health. Health Psychol. 2018;37(12):1081-1091.
- 28. Elder JP, Ayala GX, Parra-Medina D, Talavera GA. Health communication in the Latino community: issues and approaches. Annu Rev Public Health. 2009;30:227-251.
- 29. Ayala GX, Vaz L, Earp JA, Elder JP, Cherrington A. Outcome effectiveness of the lay health advisor model among Latinos in the United States: an examination by role. Health Educ Res. 2010;25(5):815-840.

- 30. Orsmond GI, Cohn ES. The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions. OTJR (Thorofare N J). 2015;35(3):169-177.
- 31. Pena MM, Dixon B, Taveras EM. Are you talking to ME? The importance of ethnicity and culture in childhood obesity prevention and management. Childhood obesity (Print). 2012;8(1):23-27.
- 32. U. S. Census Bureau. American Community Survey. Author. https://www.census.gov/programs-surveys/acs/data.html. Published 2013. Accessed.
- 33. Singh GK, Siahpush M, Kogan MD. Rising social inequalities in US childhood obesity, 2003-2007. Ann Epidemiol. 2010;20(1):40-52.
- 34. Biener AI, Cawley J, Meyerhoefer C. The Medical Care Costs of Youth Obesity: An Instrumental Variables Approach. National Bureau of Economic Research;2017.
- 35. Bolin JN, Bellamy G, Ferdinand AO, Kash BA, Helduser JW. Rural Healthy People 2020. Vol 1. College Station, TX: Texas A&M Health Science Center School of Public Health, Southwest Rural Health Research Center. http://sph.tamhsc.edu/srhrc/docs/rhp2020-volume-1.pdf; 2015.
- 36. Warne JP. Shaping the stress response: interplay of palatable food choices, glucocorticoids, insulin and abdominal obesity. Mol Cell Endocrinol. 2009;300(1-2):137-146.
- 37. Gutman LM MVTT, . Financial strain, neighborhood stress, parenting behaviors, and adolescent adjust ment in urban African-American families. J Res Adolesc. 2005;15:425–449.
- 38. van Jaarsveld CH, Fidler JA, Steptoe A, Boniface D, Wardle J. Perceived stress and weight gain in adolescence: a longitudinal analysis. Obesity (Silver Spring, Md). 2009;17(12):2155-2161.
- 39. Lissau I, Sorensen TI. Parental neglect during childhood and increased risk of obesity in young adulthood. Lancet. 1994;343(8893):324-327.
- 40. Hughes SO, Power TG, Liu Y, Sharp C, Nicklas TA. Parent emotional distress and feeding styles in low-income families. The role of parent depression and parenting stress. Appetite. 2015;92:337-342.
- 41. Urizar GG, Hurtz SQ, Ahn DK, King AC, Albright CL, Atienza AA. Influence of maternal stress on successful participation in a physical activity intervention: the IMPACT Project. Women Health. 2005;42(4):63-82.
- 42. Dallman MF, Pecoraro N, Akana SF, et al. Chronic stress and obesity: a new view of "comfort food". Proc Natl Acad Sci U S A. 2003;100(20):11696-11701.
- 43. Romero AJ. A pilot test of the Latin active hip hop intervention to increase physical activity among low-income Mexican-American adolescents. Am J Health Promot. 2012;26(4):208-211.
- 44. Olvera N, Bush JA, Sharma SV, Knox BB, Scherer RL, Butte NF. BOUNCE: a community-based mother–daughter healthy lifestyle intervention for low-income Latino families. Obesity. 2010;18(S1):S102-S104.
- 45. Barkin SL, Gesell SB, Poe EK, Ip EH. Changing overweight Latino preadolescent body mass index: the effect of the parent-child dyad. Clin Pediatr. 2011;50(1):29-36.
- 46. Summerbell CD, Waters E, Edmunds L, Kelly S, Brown T, Campbell KJ. Interventions for preventing obesity in children. The Cochrane database of systematic reviews. 2005;3(3).

- 47. Skelton JA, Buehler C, Irby MB, Grzywacz JG. Where are family theories in family-based obesity treatment?: conceptualizing the study of families in pediatric weight management. Int J Obes (Lond). 2012;36(7):891-900.
- 48. Sosa ET. Mexican American mothers' perceptions of childhood obesity: a theory-guided systematic literature review. Health Educ Behav. 2012;39(4):396-404.
- 49. Haldeman LA, Gruber KJ, Ingram KP. Determinants of food security and diet among rural and urban latino/hispanic immigrants. J Hunger Environ Nutr. 2008;2(4):67-83.
- 50. Allen ML, Elliott MN, Morales LS, Diamant AL, Hambarsoomian K, Schuster MA. Adolescent participation in preventive health behaviors, physical activity, and nutrition: differences across immigrant generations for Asians and Latinos compared with Whites. Am J Public Health. 2007;97(2):337-343.
- 51. Sussner KM, Lindsay AC, Greaney ML, Peterson KE. The influence of immigrant status and acculturation on the development of overweight in Latino families: a qualitative study. Journal of immigrant and minority health / Center for Minority Public Health. 2008;10(6):497-505.
- 52. Popkin BM, Udry JR. Adolescent obesity increases significantly in second and third generation U.S. immigrants: the National Longitudinal Study of Adolescent Health. J Nutr. 1998;128(4):701-706.
- 53. Martinez SM, Rhee K, Blanco E, Boutelle K. Maternal attitudes and behaviors regarding feeding practices in elementary school-aged Latino children: a pilot qualitative study on the impact of the cultural role of mothers in the US-Mexican border region of San Diego, California. J Acad Nutr Diet. 2014;114(2):230-237.
- 54. Lindsay AC, Sussner KM, Greaney ML, Peterson KE. Latina mothers' beliefs and practices related to weight status, feeding, and the development of child overweight. Public Health Nurs. 2011;28(2):107-118.
- 55. Baughcum AE, Burklow KA, Deeks CM, Powers SW, Whitaker RC. Maternal feeding practices and childhood obesity: a focus group study of low-income mothers. Arch Pediatr Adolesc Med. 1998;152(10):1010-1014.
- 56. Reifsnider E, Flores-Vela AR, Beckman-Mendez D, Nguyen H, Keller C, Dowdall-Smith S. Perceptions of children's body sizes among mothers living on the Texas-Mexico border (La Frontera). Public Health Nurs. 2006;23(6):488-495.
- 57. Del Parigi A. Neuroanatomical correlates of hunger and satiety in lean and obese individuals. In: Dube L, Bechara A, Dagher A, et al., eds. Obesity Prevention. Academic Press; 2010:253-271
- 58. Shonkoff ET, Dunton GF, Chou CP, Leventhal AM, Bluthenthal R, Pentz MA. Direct and indirect effects of parent stress on child obesity risk and added sugar intake in a sample of Southern California adolescents. Public Health Nutr. 2017;20(18):3285-3294.
- 59. Nyklicek I, Mommersteeg PM, Van Beugen S, Ramakers C, Van Boxtel GJ. Mindfulness-based stress reduction and physiological activity during acute stress: a randomized controlled trial. Health Psychol. 2013;32(10):1110-1113.
- 60. Coatsworth JD, Duncan LG, Nix RL, et al. Integrating mindfulness with parent training: effects of the Mindfulness-Enhanced Strengthening Families Program. Dev Psychol. 2015;51(1):26-35.
- 61. Olson KL, Emery CF. Mindfulness and weight loss: a systematic review. Psychosom Med. 2015;77(1):59-67.

- 62. Rogers JM, Ferrari M, Mosely K, Lang CP, Brennan L. Mindfulness-based interventions for adults who are overweight or obese: a meta-analysis of physical and psychological health outcomes. Obes Rev. 2017;18(1):51-67.
- 63. Kristeller JL, Wolever RQ. Mindfulness-based eating awareness training for treating binge eating disorder: the conceptual foundation. Eating disorders. 2011;19(1):49-61.
- 64. Dumas JE. Mindfulness-based parent training: strategies to lessen the grip of automaticity in families with disruptive children. J Clin Child Adolesc Psychol. 2005;34(4):779-791.
- 65. Halperin DT, Laux J, LeFranc-Garcia C, Araujo C, Palacios C. Findings From a Randomized Trial of Weight Gain Prevention Among Overweight Puerto Rican Young Adults. J Nutr Educ Behav. 2018.
- Kabat-Zinn J. Mindfulness-based interventions in context: past, present, and future. Clinical psychology:Science and practice. 2003;10(2):144–156.
- 67. Coatsworth JD, Duncan LG, Greenberg MT, Nix RL. Changing Parent's Mindfulness, Child Management Skills and Relationship Quality With Their Youth: Results From a Randomized Pilot Intervention Trial. Journal of child and family studies. 2010;19(2):203-217.
- 68. Duncan LG, Coatsworth JD, Greenberg MT. A model of mindful parenting: implications for parent-child relationships and prevention research. Clin Child Fam Psychol Rev. 2009;12(3):255-270.
- 69. Jastreboff AM, Chaplin TM, Finnie S, et al. Preventing Childhood Obesity Through a Mindfulness-Based Parent Stress Intervention: A Randomized Pilot Study. J Pediatr. 2018;202:136-142.e131.
- 70. Dahmer S. Do you have any advice on how to help with this problem of access to CAM therapies for patients without financial resources? Explore (NY). 2007;3(5):546.
- 71. Hernandez R, Garcia J, Stern M. Teens Tracking 4 Health (TT4H): a school-based weight intervention utilizing real-time tracking technology. Paper presented at American School Health Conference; 2015, October.
- 72. Stern M, Lamanna J, C. R, et al. Adaptation of an obesity intervention program for pediatric cancer survivors (NOURISH-T). Clin Pract Pediatr Psychol. 2013;1(3):264-275.
- 73. Stern M, Ewing L, Davila E, Thompson AL, Hale G, Mazzeo S. Design and rationale for NOURISH-T: a randomized control trial targeting parents of overweight children off cancer treatment. Contemp Clin Trials. 2015;41:227-237.
- 74. Mazzeo SE, Kelly NR, Stern M, et al. Nourishing Our Understanding of Role Modeling to Improve Support and Health (NOURISH): design and methods. Contemp Clin Trials. 2012;33(3):515-522.
- 75. Mazzeo SE, Kelly NR, Stern M, et al. Parent skills training to enhance weight loss in overweight children: evaluation of NOURISH. Eat Behav. 2014;15(2):225-229.
- 76. Stern M, Mazzeo S, Porter J, Gerke C, Bryan D, Laver J. Self-esteem, teasing and quality of life: African American adolescent girls participating in a family-based pediatric overweight intervention. J Clin Psychol Med Settings. 2006;13(3):217-228.

- 77. Whitlock EP, O'Connor EA, Williams SB, Beil TL, Lutz KW. Effectiveness of weight management interventions in children: a targeted systematic review for the USPSTF. Pediatrics. 2010;125(2):e396-418.
- 78. Skelton JA, Beech BM. Attrition in paediatric weight management: a review of the literature and new directions. Obes Rev. 2011;12(5):e273-281.
- 79. Perez LG, Arredondo EM, Elder JP, Barquera S, Nagle B, Holub CK. Evidence-based obesity treatment interventions for Latino adults in the U.S.: a systematic review. Am J Prev Med. 2013;44(5):550-560.
- 80. Bean MK, Wilson DB, Thornton LM, Kelly N, Mazzeo SE. Dietary intake in a randomized-controlled pilot of NOURISH: a parent intervention for overweight children. Prev Med. 2012;55(3):224-227.
- 81. Stern M, Bleck, J., Ewing, L., Davila, E., Lynn, C., Hale, G., & Mazzeo, S. NOURISH-T: Targeting Caregivers to Improve Health Behaviors in Pediatric Cancer Survivors with Obesity. Pediatric Blood and Cancer. 2018;65(10).
- 82. Rodriguez CJ, Allison M, Daviglus ML, et al. Status of cardiovascular disease and stroke in Hispanics/Latinos in the United States: a science advisory from the American Heart Association. Circulation. 2014;130(7):593-625.
- 83. Flay BR, Petraitis J. The theory of triadic influence: A new theory of health behavior with implications for preventive interventions. Adv Med Sociol. 1994;4:19-44.
- 84. Steiner-Adair C, Sjostrom L, Franko DL, et al. Primary prevention of risk factors for eating disorders in adolescent girls: learning from practice. Int J Eat Disord. 2002;32(4):401-411.
- 85. Bandura A. Social Foundations of Thought and Action. Englewood Cliffs, NJ: Prentice-Hall; 1986.
- 86. Austin SB. Prevention research in eating disorders: theory and new directions. Psychol Med. 2000;30(6):1249-1262.
- 87. Taylor SJ, Whincup PH, Hindmarsh PC, Lampe F, Odoki K, Cook DG. Performance of a new pubertal self-assessment questionnaire: a preliminary study. Paediatr Perinat Epidemiol. 2001;15(1):88-94.
- 88. Galanti GA. The Hispanic family and male-female relationships: an overview. J Transcult Nurs. 2003;14(3):180-185.
- 89. Wang JB, Cadmus-Bertram LA, Natarajan L, et al. Wearable sensor/device (Fitbit One) and SMS text-messaging prompts to increase physical activity in overweight and obese adults: A randomized controlled trial. Telemed J E Health. 2015;21(10):782-792.
- 90. Flynn MA, McNeil DA, Maloff B, et al. Reducing obesity and related chronic disease risk in children and youth: a synthesis of evidence with 'best practice' recommendations. Obes Rev. 2006;7 Suppl 1:7-66.
- 91. Campbell M, Fitzpatrick R, Haines A, et al. Framework for design and evaluation of complex interventions to improve health. Bmj. 2000;321(7262):694-696.
- 92. Castro FG, Barrera M, Jr., Martinez CR, Jr. The cultural adaptation of prevention interventions: resolving tensions between fidelity and fit. Prev Sci. 2004;5(1):41-45.
- 93. Carey MA, Asbury J. Focus group research. New York: Routledge; 2012.

- 94. Palmberg AA, Stern M, Kelly NR, et al. Adolescent girls and their mothers talk about experiences of binge and loss of control eating. Journal of child and family studies. 2014;23(8):1403-1416.
- 95. Porter, J. S., Stern M, Mazzeo SE, Evans RK, Laver J. Relations among teasing, body satisfaction, self-esteem, and depression in treatment-seeking obese African American adolescents. Journal of Black Psychology. 2013;39(4):375-395.
- 96. Stunkard, A. J., Sorensen T, Schulsinger F. Use of the Danish adoption register for the study of obesity and thinness In: S., Kety, eds. The genetics of neurological and psychiatric disorders New York, NY: Raven 1983.
- 97. Hendrickson KL, Rasmussen EB. Mindful eating reduces impulsive food choice in adolescents and adults. Health Psychol. 2017;36(3):226-235.
- 98. Levoy E, Lazaridou A, Brewer J, Fulwiler C. An exploratory study of Mindfulness Based Stress Reduction for emotional eating. Appetite. 2017;109:124-130.
- 99. Redwine LS, Henry BL, Pung MA, et al. Pilot Randomized Study of a Gratitude Journaling Intervention on Heart Rate Variability and Inflammatory Biomarkers in Patients With Stage B Heart Failure. Psychosom Med. 2016;78(6):667-676.
- 100. Redwine LS, Tsuang M, Rusiewicz A, et al. A pilot study exploring the effects of a 12-week t'ai chi intervention on somatic symptoms of depression in patients with heart failure. J Altern Complement Med. 2012;18(8):744-748.
- 101. Linke SE, Noble M, Hurst S, et al. An Exercise-Based Program for Veterans with Substance Use Disorders: Formative Research. J Psychoactive Drugs. 2015;47(3):248-257.
- 102. Wilson KL, Tomfohr L, Edwards K, et al. Effects of Aerobic Fitness and Adiposity on Coagulation Biomarkers in Men vs. Women with Elevated Blood Pressure. The European journal of cardiovascular medicine. 2012;2(2):122.
- 103. Ammerman A, Leung MM, Cavallo D. Addressing disparities in the obesity epidemic. N C Med J. 2006;67(4):301-304.
- 104. Stewart DA, Carter JC, Drinkwater J, Hainsworth J, Fairburn CG. Modification of eating attitudes and behavior in adolescent girls: a controlled study. Int J Eat Disord. 2001;29(2):107-118.
- 105. Bracero W. Intimidades: confianza, gender, and hierarchy in the construction of Latino-Latina therapeutic relationships. Cult Divers Ment Health. 1998;4(4):264-277.
- 106. U.S. Department of Health and Human Services NIoH NH, Lung and Blood Institute,. Families finding the balance: A parent handbook. (NIH Publication No. 05-5273). http://www.nhlbi.nih.gov/health/educational/wecan/tools-resources/nutrition.htm. Published 2005. Accessed October 4, 2014.
- 107. Lescano CM, Brown LK, Raffaelli M, Lima LA. Cultural factors and family-based HIV prevention intervention for Latino youth. J Pediatr Psychol. 2009;34(10):1041-1052.
- 108. Lescano C, Calcano E, Mayor M, Porter M, Marhefka S, Brown L. A randomized controlled trial of a family-based HIV prevention intervention for Latino parent-adolescent dyads, Manuscript in preparation, 2019.
- 109. Koskan A, Friedman DB, Messias DK, Brandt HM, Walsemann K. Sustainability of promotora initiatives: program planners' perspectives. J Public Health Manag Pract. 2013;19(5):E1-9.

110. London L, Hurtado-de-Mendoza A, Song M, Nagirimadugu A, Luta G, Sheppard VB. Motivators and barriers to Latinas' participation in clinical trials: the role of contextual factors. Contemp Clin Trials. 2015;40:74-80.